CLINICAL TRIAL: NCT02303106
Title: Interaction Between Paracetamol and Lamotrigine: A Clinical Interaction Study.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Per Damkier (Other)
Responsible Party: Sponsor-Investigator, Per Damkier, Head Consultant, MD, Ph.D., Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-386
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: AUC exposure to lamotrigine
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lamotrigine (Active Comparator): lamotrigine alone
  Interventions: Drug: Lamotrigine
- Lamotrigine + paracetamol (Experimental): Lamotrigine + paracetamol
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine

SUMMARY:
The investigators will study the effect of paracetamol on the steady state metabolism of lamotrigine in 12 healthy male volunteers.

Subjects will receive lamotrigine, slowly titrated from 25 mg daily to 100 mg daily over 28 days. On day 36, full plasma and urine PK samples will be drawn. On days 37-40 the subject will be co-administered 1 gr paracetamol 4 times daily. On day 40 the sampling will be repeated.

Primary outcome parameter is Lamotrigine AUC before and after coadministration of paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy no medication use
* Informed consent

Exclusion Criteria:

* Allergy to paracetamol or lamotrigine

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Lamotrigine AUC | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, MD, Principal Investigator — Head Consultant Clinical Pharmacology
Locations (1):
- University of Southern Denmark, Odense, Denmark